CLINICAL TRIAL: NCT07284849
Title: A Randomized, Double-Blind, Phase 3 Study of Standard-of-Care Chemotherapy and Bevacizumab With or Without INCA33890 in the First-Line Treatment of Metastatic Microsatellite Stable Colorectal Cancer
Brief Title: A Study to Evaluate the Efficacy and Safety of Standard-of-Care Chemotherapy and Bevacizumab With or Without INCA33890 in the First-Line Treatment of Metastatic Microsatellite Stable Colorectal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCA033890-303; 2025-523735-19-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2025-12-09; First posted 2025-12-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: CRC (Colorectal Cancer)
Keywords: Metastatic Colorectal Cancer; Colon Cancer; INCA33890
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Bevacizumab; Folfox protocol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- INCA33890 (Experimental): INCA33890 will be administered in combination with bevacizumab and FOLFOX at the protocol-defined dose.
  Interventions: Drug: INCA33890; Drug: Bevacizumab; Drug: FOLFOX
- Placebo (Placebo Comparator): Placebo will be administered in combination with bevacizumab and FOLFOX at the protocol-defined dose.
  Interventions: Drug: Placebo; Drug: Bevacizumab; Drug: FOLFOX

INTERVENTIONS:
Drug: INCA33890 — INCA33890 will be administered at protocol defined dose.
  Arms: INCA33890
Drug: Placebo — Placebo will be administered at protocol defined dose.
  Arms: Placebo
Drug: Bevacizumab — Bevacizumab will be administered at protocol defined dose.
Drug: FOLFOX — FOLFOX will be administered at protocol defined dose.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of standard-of-care chemotherapy and bevacizumab with or without INCA33890 in the first-line treatment of metastatic microsatellite stable colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV colorectal adenocarcinoma not amenable to curative resection.
* No prior systemic treatment for unresectable or metastatic disease. Participants who received adjuvant or neoadjuvant therapy may enroll if there was no recurrence within 12 months of the end of treatment.
* Measurable disease per RECIST v1.1.
* ECOG performance status of 0 or 1.
* Adequate organ function determined by laboratory results.

Exclusion Criteria:

* MSI-H/dMMR per historical data in the medical record.
* BRAF V600E mutation per historical data in the medical record.
* Untreated and/or progressing CNS metastases.
* History of other malignancy within 2 years.
* Treatment with an anti-PD-(L)1 or other immune checkpoint inhibitor for any indication within the last 3 years.
* Active autoimmune disease that has required systemic treatment in the past 2 years.
* Significant concurrent and/or uncontrolled medical condition.
* History of organ transplant, including allogeneic stem cell transplantation.

Other protocol-defined inclusion/exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2028-12-29 (Estimated); Study Completion 2029-09-28 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 3 years
  Defined as the time from the date of randomization to the date of the first documented progression as determined by the investigator per Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 4 years
  Defined as the time from the date of randomization to the date of death due to any cause.
Objective response | Up to 3 years
  Defined as complete response (CR) or partial response (PR) as determined by the investigator per RECIST v1.1.
Duration of Response (DOR) | Up to 3 years
  Defined as the time from the earliest date of documented response until the earliest date of disease progression as determined by the investigator per RECIST v1.1 or death due to any cause, whichever occurs first.
Treatment Emergent Adverse Events (TEAEs) | Up to 4 years
  Adverse events reported for the first time or worsening of a pre-existing event after first dose of study treatment, up to 90 days after the last dose INCA33890/placebo (or 30 days after the last dose of any FOLFOX component or bevacizumab if later) or the start of new anticancer therapy, whichever comes first.
TEAEs leading to dose interruptions, dose reductions or discontinuation of study treatmen | Up to 4 years
  TEAEs leading to dose interruption or study drug discontinuation.
Change from baseline in EQ-5D-5L score at protocol-defined visits | Up to 4 years
  The EQ-5D-5L is a validated, self-reported instrument for assessing HRQoL across 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 response levels of severity, ranging from no problems to extreme problems. The questionnaire also includes a visual analog scale for self-rated overall health on a scale from 0 (worst imaginable health) to 100 (best imaginable health).
Change from baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-Core 30 (C30) at protocol-defined visits | Up to 4 years
  The EORTC QLQ-C30 is a validated, self-administered questionnaire developed to assess the quality of life in cancer patients. It consists of 30 questions divided into several subscales, including 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, nausea and vomiting, and pain), a global health status/QoL scale, and a number of single-item measures that assess additional symptoms such as dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties.
Change from baseline in Functional Assessment of Cancer Therapy Colorectal Symptom Index (FCSI)-9 score at protocol-defined visits | Up to 4 years
  The FCSI-9 is a 9-item questionnaire derived from the FACT-C questionnaire to be a briefer, more targeted symptom-specific measure for patients with CRC. The FCSI-9 assesses common symptoms of CRC, including energy, pain, weight loss, nausea, diarrhea, swelling or cramps in the stomach area, appetite, ability to enjoy life, and overall quality of life. The questionnaire is scored to produce a single total score, with a higher score indicating less symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (197):
- United States (49):
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Providence Medical Foundation, Fullerton, California
  - University of California Los Angeles Health, Los Angeles, California
  - Hartford Hospital, Hartford, Connecticut
  - University of Florida Health, Gainesville, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Advent Health, Orlando, Florida
  - Orlando Health Cancer Institute Downtown Orlando, Orlando, Florida
  - Ascension Sacred Heart Pensacola, Pensacola, Florida
  - St Lukes Mountain States Tumor Institute Msti Boise, Boise, Idaho
  - Endeavor Health, Evanston, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Community Health Network, Indianapolis, Indiana
  - Saint Agnes Hospital, Baltimore, Maryland
  - Cancer Center For Blood Disorders A Division of American Oncology Partners P.A, Bethesda, Maryland
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint Luke'S Hospital of Kansas City, Kansas City, Missouri
  - Midamerica Cancer Care, Kansas City, Missouri
  - Oncology Hematology Associates, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Morristown Medical Center, Morristown, New Jersey
  - Icahn School of Medicine At Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ny Cancer and Blood Specialists, Patchogue, New York
  - University of Rochester, Rochester, New York
  - Montefiore Einstein For Cancer Care, The Bronx, New York
  - Messino Cancer Center, Asheville, North Carolina
  - The University of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - Ohio State University-Arthur G James Comprehensive Cancer Center, Columbus, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital Cancer Institute, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center Upmc Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Cancer Care Associates of York, York, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Provision Center For Biomedical Research, Knoxville, Tennessee
  - Sarah Cannon Research Institute Scri Oncology Partners, Nashville, Tennessee
  - Shivers Cancer Center, Austin, Texas
  - Texas Oncology, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Md Anderson Cancer Center, Houston, Texas
  - Shenandoah Oncology, Winchester, Virginia
  - Vandalia Health Charleston Area Medical Center, Charleston, West Virginia
  - West Virginia University, Morgantown, West Virginia
- Argentina (10):
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - Investigaciones Clinicas Moleculares Icm, Buenos Aires
  - Instituto Medico Especializado Alexander Fleming, Buenos Aires
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Instituto de Investigaciones Clinicas Cordoba S.A., Córdoba
  - Hospital Privado Centro Medico de Cordoba S.A, Córdoba
  - Centro Oncologico Riojano Integral (Cori), La Rioja
  - Investigaciones Oncologicas C Colon, Mar del Plata
  - Instituto de Oncologia de Rosario, Rosario
  - Exelsus Srl, San Miguel de Tucumán
- Australia (13):
  - Border Cancer Hospital Dispensary - Albury Wodonga Regional Cancer Centre, Albury, New South Wales
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Prince of Wales Hospital Au, Randwick, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Wollongong Hospital, Wollongong, New South Wales
  - Townsville Cancer Centre, Townsville, Queensland
  - Princess Alexandra Hospital Australia, Woolloongabba, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch
- Austria (4):
  - Lkh - Universitaetsklinikum Graz, Graz
  - Ordensklinikum Krankenhaus Der Barmherzigen Schwestern Linz, Linz
  - Lkh - Universitatsklinikum Der Pmu Salzburg, Salzburg
  - Akh - Medizinische Universität Wien, Vienna
- Belgium (6):
  - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires Ucl Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen (Uza), Edegem
  - Universitair Ziekenhuis Gent (Uz Gent), Ghent
  - Universitaire Ziekenhuis Leuven - Gasthuisberg, Leuven
  - Chu Ucl Namur University Hospital Mont-Godinne, Yvoir
- Brazil (13):
  - Fundacao Pio Xii Hospital de Cancer de Barretos, Barretos
  - Centro de Pesquisas Clinica Reichow, Blumenau
  - Oncosite - Centro de Pesquisa Clinica E Oncologia, Ijuí
  - Clinica de Neoplasias Litoral Ltda, Itajaí
  - Liga Norte-Rio-Grandense Contra O Câncer, Natal
  - Irmandade Da Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
  - Centro Gaucho Integrado de Oncologia, Hematologia, Ensino E Pesquisa - Hospital Mae de Deus, Porto Alegre
  - Hospital Das Clínicas Fmrp-Usp, Ribeirão Preto
  - Nob - Nucleo de Oncologia Da Bahia, Salvador
  - Cepho - Centro de Estudos E Pesquisas de Hematologia E Oncologia, Santo André
  - Fundacao Faculdade Regional de Medicina de Sao Jose Do Rio Preto, SAO JOSE RIO Preto
  - Icavc - Instituto Do Câncer Arnaldo Vieira de Carvalho, São Paulo
- Canada (5):
  - Cross Cancer Institute, Edmonton, Alberta
  - Southlake Regional Health Center, Newmarket, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Hôtel-Dieu de Lévis, Lévis, Quebec
  - McGill University Health Centre Research Institute, Montreal, Quebec
- Denmark (4):
  - Aalborg Universitetshospital, Aalborg
  - OUH, Odense C
  - Sjaellands Universitetshospital, Roskilde
  - Sygehus Lillebælt - Vejle, Vejle
- France (10):
  - Chu Bordeaux-Hopital Pellegrin, Bordeaux
  - Institut Paoli Calmettes, Marseille
  - Hôpital de La Timone, Marseille
  - Hospital Universitaire Pitie-Salpetriere, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hospital de La Miletrie, Poitiers
  - Chu de Reims, Reims
  - University Hospital of Saint Etienne, Saint-Etienne
  - Chu Toulouse Hopital Rangueil, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (13):
  - Charite - Campus Virchow-Klinikum, Berlin
  - University Hospital Carl Gustav Carus, Dresden
  - Universitaetsklinikum Essen, Essen
  - Krankenhaus Nordwest Gmbh, Frankfurt am Main
  - University Medical Center Freiburg, Freiburg im Breisgau
  - University Medical Centre Hamburg-Eppendorf Centre of Oncology, Hamburg
  - Asklepios Tumorzentrum Hamburg, Hamburg
  - Hannover Medical School, Hanover
  - Uksh Campus Lubeck, Lübeck
  - Klinikum Der University Munchen - Campus Grosshadern, München
  - Klinikum Neuperlach, München
  - Universitaetsklinikum Regensburg, Regensburg
  - Universitatkinikums Ulm, Ulm
- Italy (16):
  - Azienda Ospedaliero Universitaria Delle Marche, Ancona
  - Irccs Centro Di Riferimento Oncologico, Aviano
  - Istituto Tumori Giovanni Paolo Ii Irccs Ospedale Oncologico Bari, Bari
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia
  - Istituto Di Candiolo Fondazione Del Piemonte Per L'Oncologia - Irccs, Candiolo
  - Comitato Etico Fondazione Irccs Istituto Nazionale Dei Tumori Milano, Milan
  - Asst Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera Universitaria- Università Degli Studi Della Campania "Luigi Vanvitelli", Napoli
  - Iov - Istituto Oncologico Veneto Irccs, Padua
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Ospedale Santa Maria Delle Croci, Ravenna
  - Arcispedale S. Maria Nuova Azienda Ospedaliera Di Reggio Emilia, Reggio Emilia
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Irccs Istituto Clinico Humanitas, Rozzano
  - I.R.C.C.S. Casa Sollievo Della Sofferenza, San Giovanni Rotondo
  - Centro Ricerche Cliniche Di Verona, Verona
- Japan (11):
  - Chiba Cancer Center, Chiba
  - National Cancer Center Hospital, Chūōku
  - Nho Kyushu Cancer Center, Fukuoka
  - Saitama Medical University International Medical Center, Hidaka-shi
  - National Cancer Center Hospital East, Kashiwa-shi
  - Cancer Institute Hospital of Jfcr, Kōtoku
  - Nho Shikoku Cancer Center, Matsuyama
  - Osaka International Cancer Institute, Osaka
  - The University of Osaka Hospital, Suita-shi
  - Shizuoka Cancer Center, Sunto-gun
  - Kanagawa Cancer Center, Yokohama
- Netherlands (4):
  - Meander Medisch Centrum, Amersfoort
  - Martini Ziekenhuis, Groningen
  - Maastricht Umc+, Maastricht
  - Erasmus Medical Center, Rotterdam
- Norway (3):
  - Haukeland Universitetssjukehus, Bergen
  - Akershus Universitetssykehus Hf, Lørenskog
  - Oslo Universitetssykehus, Oslo
- Poland (4):
  - Wojewodzkie Centrum Szpitalne Kotliny Jeleniogorskiej, Jelenia Góra
  - Mazowiecki Szpital Wojewodzki Im. SW. Jana Pawla Ii W Siedlcach Sp Z O O, Siedlce
  - Luxmed Onkologia Sp. Z O.O., Warsaw
  - Narodowy Instytut Onkologii Im. Marii Skłodowskiej-Curie - Państwowy Instytut Badawczy, Warsaw
- Pan American Center For Oncology Trials Llc Dorado Office, Dorado, Puerto Rico
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - The Catholic University of Korea Seoul St. Mary'S Hospital, Seoul
- Spain (15):
  - Hospital Universitari Germans Trias I Pujol, Badalona
  - Hospital General Universitario Vall D Hebron, Barcelona
  - Hospital Clinic Barcelona Main, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Complejo Hospitalario Universitario Insular-Materno Infantil, Las Palmas de Gran Canaria
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda
  - Son Espases University Hospital, Palma de Mallorca
  - Hospital Universitario de Navarra, Pamplona
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitari Mutua de Terrassa, Terrassa
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Switzerland (3):
  - Inselspital - Universitaetsspital Bern, Bern
  - Chuv, Lausanne University Hospital, Lausanne
  - Hoch Health Ostschweiz, Sankt Gallen
- United Kingdom (8):
  - Bristol Haematology and Oncology Centre, Bristol
  - Velindre Cancer Centre, Cardiff
  - St James University Hospital, Leeds
  - Barts Hospital, London
  - Guys Hospital, London
  - Kent Oncology Centre - Maidstone Hospital, Maidstone
  - The Christie Nhs Foundation Trust Uk, Manchester
  - The Royal Marsden Nhs Foundation Trust - Chelsea, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: A Study to Evaluate the Efficacy and Safety of Standard-of-Care Chemotherapy and Bevacizumab With or Without INCA33890 in the First-Line Treatment of Metastatic Microsatellite Stable Colorectal Cancer — https://incyteclinicaltrials.com/studies/nct07284849